CLINICAL TRIAL: NCT00982397
Title: The PainFree SST Clinical Study: Clinical Study to Evaluate System Safety and Clinical Performance of the Protecta ICD + CRT-D and to Assess the Capacity of the Protecta Features to Reduce Inappropriate Shocks.
Brief Title: Safety and Clinical Performance of the Protecta ICD and CRT-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PainFree SST
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Tachyarrhythmias; Heart Failure; Ventricular Dysfunction
MeSH Terms: conditions — Tachycardia; Heart Failure; Ventricular Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-chamber detetction (Experimental): Patients implanted with a Protecta VR-ICD.
  Interventions: Device: Protecta VR-ICD
- Dual-chamber detection (Experimental): Patients implanted with a Protecta DR-ICD or CRT-D.
  Interventions: Device: Protecta DR-ICD or CRT-D

INTERVENTIONS:
Device: Protecta VR-ICD — Protecta single-chamber implantable cardioverter defibrillators.
  Arms: Single-chamber detetction
Device: Protecta DR-ICD or CRT-D — Protecta dual-chamber implantable cardioverter defibrillators and cardiac resynchronization therapy defibrillators.
  Arms: Dual-chamber detection

SUMMARY:
The purpose of the study is two-fold. In Phase I (Protecta Clinical Study), system performance will be evaluated. In Phase II (PainFree SST), the inappropriate shock-free rate at one year of subjects implanted with a Medtronic Protecta implantable cardioverter defibrillator (ICD) and cardiac resynchronization therapy defibrillator (CRT-D) will be evaluated.

DETAILED DESCRIPTION:
The PainFree SST study was a prospective, multicenter clinical trial, which was conducted in two consecutive phases. Phase I assessed safety as determined by assessment of delays in ventricular fibrillation (VF) arrhythmia detection time using new algorithms. Phase II assessed the influence of new algorithms on inappropriate and unnecessary shocks at 1 year of follow-up. Subjects enrolled in Phase I continued in Phase II of the study and data from all enrolled subjects contributed to the analysis of Phase II objectives. A sub-study of Phase II randomized secondary prevention subjects to either 18/24 NID or 30/40 NID in order to assess the safety of prolonged detection in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting one of the following criteria can be included in Phase I of the study:

  * Patients indicated (per local indications) for a dual chamber implantable cardioverter defibrillator (DR-ICD)/cardiac resynchronization therapy defibrillator (CRT-D)
  * Patients undergoing a device replacement or upgrade to DR-ICD or CRT-D and with the protocol required leads (patients must be enrolled prior to implant)
* Patients meeting one of the following criteria can be included in Phase II of the study:

  * Patients indicated for a DR-ICD/VR-ICD/CRT-D device and intended to receive a Protecta device
  * Patients undergoing a DR-ICD/VR-ICD/CRT-D device replacement or an upgrade to a Protecta DR-ICD/VR-ICD or CRT-D
  * Patients indicated for a DR-ICD/VR-ICD/CRT-D already implanted with a Protecta device and the protocol required leads, who have not yet been discharged after implant

Exclusion Criteria:

* Patients with a mechanical tricuspid heart valve
* Patients enrolled or intended to participate in any concurrent drug and/or device study, which would confound the results of this trial as determined by Medtronic, during the course of this clinical study
* Patients with medical conditions that preclude the testing required for all patients by the study protocol or that otherwise limit study participation required for all patients
* Patients with exclusion criteria required by local law (e.g. age, pregnancy, breast feeding, etc)
* Patients anticipated not being able to complete the study
* Patients unwilling to provide written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2770 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Meijer, Dr., Principal Investigator — Eindhoven, The Netherlands; A. Auricchio, Prof., Principal Investigator — Lugano, Switzerland; T. Kurita, Dr., Principal Investigator — Higashi-Osaka, Japan; E.J. Schloss, Dr., Principal Investigator — Cincinnati Ohio, USA; L. Sterns, Dr., Principal Investigator — Victoria, British Columbia, Canada
Locations (122):
- United States (29):
  - Birmingham Heart Clinic PC, Birmingham, Alabama
  - CardioVasular Associates of Mesa, Mesa, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - LA Cardiology Associates, Los Angeles, California
  - Cardiology Consultants of Napa Valley, Napa, California
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida Health at Jacksonville, Jacksonville, Florida
  - Arrhythmia Syncope Consultants LLC, Miami, Florida
  - Indiana Heart Physicians, Indianapolis, Indiana
  - Cardiovascular Research of Northwest Indiana, Munster, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Delmarva Heart Research Foundation, Salisbury, Maryland
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - Saint John's Medical Research Inc, Springfield, Missouri
  - Saint Louis Heart & Vascular PC, St Louis, Missouri
  - Cardiology PC, Syracuse, New York
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Ohio Heart and Vascular, Cincinnati, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Central Bucks Cardiology, Doylestown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Pee Dee Cardiology, Florence, South Carolina
  - Cardiology Consultants PA, Spartanburg, South Carolina
  - Centennial Heart Cardiovascular Consultants LLC, Nashville, Tennessee
  - Hall-Garcia Cardiology Associates, Houston, Texas
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Spokane Cardiology, Spokane, Washington
  - Columbia St. Mary's Hospital, Milwaukee, Wisconsin
- Austria (3):
  - LKH - Universitätsklinikum Graz, Graz
  - Landesklinikum St. Pölten, Sankt Pölten
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Canada (10):
  - Saint Paul's Hospital (Vancouver BC), Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Institut Universitaire de Cardiologieet de Pneumologie de Québec (IUCPQ), Halifax, Nova Scotia
  - Newmarket Electrophysiology Research Group, Newmarket, Ontario
  - Queen Elizabeth II Health Sciences Centre, Halifax
  - Kelowna Arrhythmia Research, Kelowna
  - Queen's University & Kingston General Hospital, Kingston
  - London Health Sciences Centre - University Campus, London
  - Montreal Heart Institute, Montreal
  - University of Ottawa Heart Institute, Ottawa
- Colombia (3):
  - Fundacion Cardioinfantil, Bogotá
  - Hospital Cardiovascular del Nino, Bogotá
  - Clinica Cardiovascular Santa Maria, Medellín
- Krajska nemocnice Liberec a.s. - Kardiocentrum, Liberec, Czechia
- Denmark (2):
  - Aalborg Sygehus, Aalborg
  - Aarhus Universitetshospital - Skejby, Aarhus
- Germany (20):
  - Herz- und Gefässzentrum Bad Bevensen, Bad Bevensen
  - Herz- und Diabeteszentrum NRW - Ruhr-Universität Bochum, Bad Oeynhausen
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Berufsgenossenschaftliche Universitätsklinik Bergmannsheil GmbH, Bochum
  - Universitätsklinikum Bonn, Bonn
  - MVZ am Küchwald GmbH ambulantes Herz Zentrum Chemnitz, Chemnitz
  - Klinikum Coburg GmbH, Coburg
  - Kardiocentrum Frankfurt an der Klinik Rotes Kreuz, Frankfurt
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Ruprecht-Karls-Universität, Heidelberg
  - Westpfalz-Klinikum GmbH - Standort I Kaiserslautern, Kaiserslautern
  - Herz Zentrum Bodensee, Konstanz
  - Klinikum Ludwigsburg - Akademisches Lehrkrankenhaus der Universität Heidelberg, Ludwigsburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Städtische Kliniken München GmbH - Klinikum Bogenhausen, München
  - Städtische Kliniken Neuss Lukaskrankenhaus GmbH-Akad.Lehrkrankenhaus d. Heinrich-Heine-Universität, Neuss
  - Universitätsmedizin Rostock, Rostock
  - Herz- und Kreislaufzentrum Rotenburg a.d. Fulda GmbH, Rotenburg A.d. Fulda
  - Asklepios Kliniken Schwalm - Eder GmbH - Klinikum Schwalmstadt, Schwalmstadt
  - Heinrich-Braun-Klinikum Zwickau gemeinnützige GmbH, Zwickau
- India (2):
  - Care Institute of Medical Sciences, Ahmedabad
  - Medanta-The Medicity, Gūrgaon
- Israel (9):
  - Barzilai Medical Center Ashkelon, Ashkelon
  - Soroka University Medical Center, Be'er Sheba
  - Carmel Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Ospedale classificato ed equiparato Sacro Cuore - Don Calabria, Negrar
  - Azienda Complesso Ospedaliero San Filippo Neri - Ospedale San Filippo Neri, Rome
- Japan (14):
  - Hirosaki University School of Medicine & Hospital, Hirosaki, Aomori
  - Kansai Rosai Hospital, Amagasak, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Kinki University Hospital, Osakasaya, Osaka
  - National Cerebral and Cardiovasuclar Center, Suita, Osaka
  - Sapporo Medical Center NTT EC, Chūōku, Sapporo
  - Akita Medical Center, Akita
  - Chiba University Hospital, Chiba
  - Kokura Memorial Hospital, Kitakyushu
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Niigata University Medical & Dental Hospital, Niigata
  - Kitasato University Hospital, Sagamihara
- Institut Jantung Negara - National Heart Institute, Kuala Lumpur, Malaysia
- Netherlands (9):
  - Medisch Centrum Alkmaar, Alkmaar
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Amphia Ziekenhuis - Locatie Molengracht Breda, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - St. Antonius Ziekenhuis, Nieuwegein
  - Universitair Medisch Centrum Utrecht, Utrecht
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Center, Riyadh
  - Prince Salman Heart Centre - King Fahad Medical City, Riyadh
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Milpark Hospital, Johannesburg, South Africa
- Spain (4):
  - Hospital De Cruces, Barakaldo
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Complejo Hospitalario Universitario de Vigo (CHUVI) - Hospital del Meixoeiro, Vigo
- Sweden (3):
  - Universitetssjukhuset i Lund, Lund
  - Universitetssjukhuset Örebro, Örebro
  - Capio S:t Görans Sjukhus, Stockholm
- Cardio Centro Ticino, Lugano, Switzerland
- Sheikh Khalifa Medical Center, Abu Dhabi, United Arab Emirates
- United Kingdom (4):
  - Royal Bournemouth Hospital, Bournemouth
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - King's College Hospital NHS Foundation Trust, London
  - Southampton General Hospital - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auricchio A, Meijer A, Kurita T, Schloss E, Brinkman K, Claessens-van Ooijen M, Sterns L. Safety, efficacy, and performance of new discrimination algorithms to reduce inappropriate and unnecessary shocks: the PainFree SST clinical study design. Europace. 2011 Oct;13(10):1484-93. doi: 10.1093/europace/eur133. Epub 2011 Jun 13. PMID 21669960
- [Result] Auricchio A, Schloss EJ, Kurita T, Meijer A, Gerritse B, Zweibel S, AlSmadi FM, Leng CT, Sterns LD; PainFree SST Investigators. Low inappropriate shock rates in patients with single- and dual/triple-chamber implantable cardioverter-defibrillators using a novel suite of detection algorithms: PainFree SST trial primary results. Heart Rhythm. 2015 May;12(5):926-36. doi: 10.1016/j.hrthm.2015.01.017. Epub 2015 Jan 28. PMID 25637563
- [Result] Sterns LD, Meine M, Kurita T, Meijer A, Auricchio A, Ando K, Leng CT, Okumura K, Sapp JL, Brown ML, Lexcen DR, Gerritse B, Schloss EJ. Extended detection time to reduce shocks is safe in secondary prevention patients: The secondary prevention substudy of PainFree SST. Heart Rhythm. 2016 Jul;13(7):1489-96. doi: 10.1016/j.hrthm.2016.03.022. Epub 2016 Mar 14. PMID 26988379
- [Result] Wollmann CG, Lawo T, Kuhlkamp V, Becker R, Garutti C, Jackson T, Brown ML, Mayr H. Implantable defibrillators with enhanced detection algorithms: detection performance and safety results from the PainFree SST study. Pacing Clin Electrophysiol. 2014 Sep;37(9):1198-209. doi: 10.1111/pace.12390. Epub 2014 Mar 25. PMID 24665992
- [Derived] Zweibel S, Cronin EM, Schloss EJ, Auricchio A, Kurita T, Sterns LD, Gerritse B, Lexcen DR, Cheng A. Estimating the incidence of atrial fibrillation in single-chamber implantable cardioverter defibrillator patients. Pacing Clin Electrophysiol. 2019 Feb;42(2):132-138. doi: 10.1111/pace.13555. Epub 2018 Dec 13. PMID 30478983
- [Derived] Kurita T, Ando K, Ueda M, Shizuta S, Okamura H, Matsumoto N, Gerritse B, Fagan DH, Schloss EJ, Meijer A, Auricchio A, Sterns LD, Okumura K; PainFree SST investigators. Comparison of ICD shock rates in Japanese and non-Japanese patients in the PainFree SST study. Pacing Clin Electrophysiol. 2018 Sep;41(9):1185-1191. doi: 10.1111/pace.13427. Epub 2018 Aug 13. PMID 29928759

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty patients were excluded from analysis, because they did not meet the eligibility criteria; 1 patient did not sign consent, 1 patient participated in a confounding trial, 8 patients did not have an implant attempted, 5 patients failed implant, and 5 patients received a device other than the Protecta.Total enrolled=2790, total analyzed=2770
Groups:
- DR-ICD/CRT-D: Patients implanted with a dual-chamber ICD (DR-ICD) or cardiac resynchronization therapy defibrillator (CRT-D).
- VR-ICD: Patients implanted with a single-chamber ICD (VR-ICD).
Period: Phase I
Arm/Group | DR-ICD/CRT-D | VR-ICD
Started | 236 | 0
Completed | 236 | 0
Not Completed | 0 | 0
Period: Phase II/Overall Study
Arm/Group | DR-ICD/CRT-D | VR-ICD
Started (Note additional subjects were enrolled for Phase II) | 2019 | 751
Secondary Prevention Randomized 18/24NID (NID=number of intervals to detect prior to therapy delivery) | 231 | 122
Secondary Prevention Randomized 30/40NID (NID=number of intervals to detect prior to therapy delivery) | 221 | 131
Completed | 2019 | 751
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DR-ICD/CRT-D | VR-ICD | Total
Number analyzed (Participants) | 2019 | 751 | 2770
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (12.1) | 61.9 (12.1) | 64.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 430 | 140 | 570
  Male | 1589 | 611 | 2200
Region of Enrollment [Number; unit: participants]
  Austria | 44 | 14 | 58
  Canada | 119 | 145 | 264
  Colombia | 18 | 4 | 22
  Czech Republic | 33 | 30 | 63
  Denmark | 60 | 42 | 102
  Germany | 248 | 57 | 305
  India | 7 | 18 | 25
  Israel | 104 | 58 | 162
  Italy | 61 | 11 | 72
  Japan | 144 | 37 | 181
  Malaysia | 17 | 2 | 19
  Netherlands | 154 | 86 | 240
  Saudi Arabia | 121 | 43 | 164
  Slovenia | 15 | 0 | 15
  South Africa | 7 | 0 | 7
  Spain | 24 | 30 | 54
  Sweden | 17 | 3 | 20
  Switzerland | 13 | 0 | 13
  United Arab Emirates | 1 | 4 | 5
  United Kingdom | 103 | 11 | 114
  United States | 709 | 156 | 865
LVEF [Mean (Standard Deviation); unit: %] | 31.8 (13.0) | 33.3 (13.5) | 32.2 (13.2)
QRS [Mean (Standard Deviation); unit: ms] | 133.7 (33.7) | 107.1 (21.9) | 125.9 (33.0)
Indication [Number; unit: participants] — Primary prevention is an ICD indication to prevent sudden cardiac death. It refers to use of ICDs in individuals who are at risk for, but have not yet had, an episode of sustained VT, VF, or cardiac arrest.
  Secondary prevention refers to an ICD indication for patients who have survived 1 or more cardiac arrests or sustained ventricular tachycardia. Patients with cardiac conditions associated with a high risk of sudden death who have unexplained syncope that is likely to be due to self-terminating ventricular arrhythmias are also considered to have a secondary prevention indication.
  participants
    Secondary Prevention | 593 | 254 | 847
    Primary Prevention | 1426 | 497 | 1923
Heart Failure Status [Number; unit: participants] — NYHA Class I-No limitation of physical activity. NYHA Class II-Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  NYHA Class III-Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  NYHA Class IV-Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  participants
    NYHA I | 232 | 187 | 419
    NYHA II | 758 | 346 | 1104
    NYHA III | 754 | 99 | 853
    NYHA IV | 30 | 8 | 38
    No Heart Failure | 245 | 109 | 354
    Unknown | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Are Inappropriate Shock Free
Description: Primary objective of Phase II. Subjects implanted with a VR device will be analyzed separately from subjects implanted with a DR / CRT-D device. An inappropriate shock is a shock delivered by the defibrillator when the patient's heart rhythm was not a tachyarrhythmia, as adjudicated by the independent Episode Review Committee .
Time Frame: Implant to one year post-implant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | DR-ICD/CRT-D | VR-ICD
Number analyzed (Participants) | 2019 | 751
percentage of patients | 98.5 [97.9 to 99.0] | 97.5 [96.1 to 98.5]
Statistical Analysis 1: Comparison: DR-ICD/CRT-D; The study was designed to include at least 1,131 patients with DR/CRT-D ICD devices in order to estimate the inappropriate shock free rate at 1 year post-implant with 1% precision; Test type: Superiority or Other; percentage of participants = 98.5, 95% CI 2-sided [97.9 to 99.0] — Therapy rates were analyzed using competing risks survival analysis methods, accounting for death as a competing risk.Therapy incidence rates were estimated using cumulative incidence functions and reported with 95% confidence interval
Statistical Analysis 2: Comparison: VR-ICD; This study was designed to include at least 610 patients with VR-ICD devices in order to estimate the inappropriate shock free rate at 1 year post-implant with a precision of 2%; Test type: Superiority or Other; percentage of participants = 97.5, 95% CI 2-sided [96.1 to 98.5] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Subjects With Unanticipated Severe Adverse Device Effects (Phase I)
Description: In Phase I, only DR-ICD/CRT-D devices were implanted, so that for Phase I objectives there is only 1 arm to report results for.
Time Frame: Implant to one month post-implant
Population: Phase I subjects (a subset of the total number of subjects) implanted with a Protecta device with at least 30 days of follow-up or a USADE within the first 30 days post-implant are included in this analysis. One hundred subjects met the criteria above and are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Phase I: Subjects enrolled in Phase I of the study (Protecta).
Arm/Group | Phase I
Number analyzed (Participants) | 100
percentage of patients | 0 [NA to 3.0] — As specified in the protocol and analysis plan, only a one-sided 95% binomial upper confidence bound is used.
Statistical Analysis 1: Comparison: Phase I; Using the one-sided one proportion Exact Test in PASS sample size software, a sample size of 76 subjects with 1-month follow-up was calculated to be required for the evaluation of this objective. To ensure adequate testing of the Protecta XT CRT-D device, the 76 subjects must have included at least 34 CRT-D subjects. Assuming an attrition rate of 10%, a sample size of 85 subjects enrolled was calculated to be required; Test type: Superiority or Other; p < 0.0001, Exact Binomial — P-value is for comparison against a performance criterion of 10%

3. Primary Outcome: Percentage of Phase I Subjects Where the Ventricular Fibrillation (VF) Detection Time With Protecta Features on is no More Than 2 Seconds Longer Than the VF Detection Time With Protecta Features Off
Description: as for outcome 2
Time Frame: At implant
Population: Of the 236 subjects implanted, 40 subjects / episodes were classified as not useable. In Phase I, only DR-ICD/CRT-D devices were implanted, so that for Phase I objectives there is only 1 arm to report results for.
Measure: Number (97.5% Confidence Interval); unit: percentage of patients
Arm/Group | Phase I
Number analyzed (Participants) | 196
percentage of patients | 100 [98.1 to NA] — As specified in the protocol and analysis plan, a one-side lower confidence bound was used.
Statistical Analysis 1: Comparison: Phase I; P, the expected proportion of successes under the null hypothesis, was 95%. α, the Type I error rate, is 0.025. Power is 90%. Pa, the assumed true proportion of successes, is 99%. Based on the above assumptions, at least 173 subjects with a useable time to VF detection testing were required for this objective. Assuming a 5% rate for the potential non-adherence to the testing protocol, the required enrollment sample size was 183; Test type: Superiority or Other; p < 0.0001, Confidence interval and hypothesis test — P-value is for comparison of the observed proportion of successes against a protocol-specified performance criterion of 95%

4. Secondary Outcome: Percentage of Secondary Prevention Subjects Who Are Syncopal Event Free
Time Frame: Implant to one year post-implant
Population: Includes randomized secondary prevention patients from Phase II.
Measure: Number; unit: percentage of patients
Groups:
- 18/24 NID: Secondary prevention subjects in Phase II randomized to 18/24 NID. (18/24 NID indicates the number of intervals used to detect VF was programmed to 18 of 24 intervals).
- 30/40 NID: Secondary prevention subjects in Phase II randomized to 30/40 NID. (30/40 NID indicates the number of intervals used to detect VF was programmed to 30 of 40 intervals).
Arm/Group | 18/24 NID | 30/40 NID
Number analyzed (Participants) | 353 | 352
percentage of patients | 96 | 96
Statistical Analysis 1: Comparison: 18/24 NID vs 30/40 NID; The expected syncopal event free rate was 0.984 in both programming groups. alpha, Type I error was 0.05. Power, 1-beta, was 80%. Non-inferiority margin 5% Based on the above assumptions and Farrington-Manning test, a total of 230 subjects was required. By further assuming 15% attrition rate and 5 % of crossover rate, a total of 300 subjects were needed; Test type: Non-Inferiority or Equivalence — Ho: p1 ≤ p2 - 0.05 Ha: p1 > p2 - 0.05 Where p1 was the syncopal event free rate at one year post implant by programming VF NID 30/40 and p2 for NID = 18/24. If the null-hypothesis was rejected it was concluded that NID = 30/40 did not decrease the syncope free rate by more than 5% compared to NID = 18/24 and hence was non-inferior; p = 0.0013, Farrington-Manning — P-Value is for non-inferiority; Risk Difference (RD) = 0.0, 90% CI 2-sided [-2.7 to 2.7] — The 90% Confidence Interval is for the difference (p1-p2), where p1=syncope free rate 30/40 arm and p2=syncope free rate 18/24 arm. Estimated value and confidence interval reflect percentages

ADVERSE EVENTS:
Time Frame: Reported Serious Adverse Events (SAEs) include events starting on or after the date of consent and through study completion, an average of 22 months.
Description: Other (non-serious) AE data were not collected for this study.
Arm/Group | DR-ICD/CRT-D | VR-ICD
Serious Adverse Events (participants affected / at risk) | 452/2019 | 125/751
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DR-ICD/CRT-D (N=2019) | VR-ICD (N=751)
Anaemia (Blood and lymphatic system disorders) | 8 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 8 | 3
Angina pectoris (Cardiac disorders) | 19 | 4
Angina unstable (Cardiac disorders) | 6 | 2
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 33 | 4
Atrial flutter (Cardiac disorders) | 10 | 2
Atrial tachycardia (Cardiac disorders) | 2 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 7 | 0
Cardiac failure (Cardiac disorders) | 108 | 29
Cardiac failure acute (Cardiac disorders) | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 4 | 0
Cardiac failure congestive (Cardiac disorders) | 6 | 2
Cardiac perforation (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 3
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Heart valve incompetence (Cardiac disorders) | 0 | 2
Hypertrophic cardiomyopathy (Cardiac disorders) | 2 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1
Mitral valve disease mixed (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 4 | 0
Palpitations (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 5 | 1
Ventricular fibrillation (Cardiac disorders) | 5 | 2
Ventricular tachyarrhythmia (Cardiac disorders) | 6 | 1
Ventricular tachycardia (Cardiac disorders) | 40 | 14
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hyperparathyroidism tertiary (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Retinopathy proliferative (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Polyp colorectal (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Adverse drug reaction (General disorders) | 0 | 2
Asthenia (General disorders) | 1 | 1
Catheter site haemorrhage (General disorders) | 1 | 0
Chest pain (General disorders) | 14 | 4
Death (General disorders) | 5 | 3
Device battery issue (General disorders) | 1 | 0
Device capturing issue (General disorders) | 1 | 0
Device dislocation (General disorders) | 32 | 3
Device electrical impedance issue (General disorders) | 2 | 0
Device extrusion (General disorders) | 1 | 0
Device failure (General disorders) | 1 | 0
Device issue (General disorders) | 1 | 0
Device lead damage (General disorders) | 9 | 2
Device lead issue (General disorders) | 3 | 3
Device malfunction (General disorders) | 1 | 0
Device misuse (General disorders) | 8 | 2
Device pacing issue (General disorders) | 5 | 0
Device stimulation issue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 2 | 0
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Implant site haematoma (General disorders) | 4 | 0
Implant site pain (General disorders) | 3 | 2
Multi-organ failure (General disorders) | 3 | 0
Oedema (General disorders) | 1 | 0
Oversensing (General disorders) | 3 | 1
Pyrexia (General disorders) | 4 | 1
Sudden cardiac death (General disorders) | 0 | 1
Undersensing (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 6 | 1
Endocarditis bacterial (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 3 | 1
Gangrene (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Implant site abscess (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 9 | 4
Infection (Infections and infestations) | 7 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Orchitis (Infections and infestations) | 1 | 0
Pleural infection (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 21 | 6
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 7 | 1
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Cardiac vein dissection (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 4 | 2
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Pocket erosion (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 4 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Arteriogram coronary (Investigations) | 4 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood pressure abnormal (Investigations) | 1 | 0
Catheterisation cardiac (Investigations) | 1 | 0
Colonoscopy (Investigations) | 0 | 1
Investigation (Investigations) | 2 | 1
Liver function test abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant non-resectable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 8 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hypokinesia (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 18 | 3
Transient ischaemic attack (Nervous system disorders) | 5 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 1
Nephritis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 4 | 0
Renal failure (Renal and urinary disorders) | 4 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 3
Renal failure chronic (Renal and urinary disorders) | 2 | 0
Renal infarct (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 3
Epiglottis ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Adrenalectomy (Surgical and medical procedures) | 1 | 0
Cardiac ablation (Surgical and medical procedures) | 1 | 0
Central venous catheter removal (Surgical and medical procedures) | 1 | 0
Corneal transplant (Surgical and medical procedures) | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Gastrectomy (Surgical and medical procedures) | 1 | 0
Heart transplant (Surgical and medical procedures) | 3 | 0
High frequency ablation (Surgical and medical procedures) | 3 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1
Indwelling catheter management (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 2 | 0
Medical device change (Surgical and medical procedures) | 11 | 0
Medical device implantation (Surgical and medical procedures) | 0 | 2
Neurostimulator implantation (Surgical and medical procedures) | 1 | 0
Radiotherapy (Surgical and medical procedures) | 0 | 1
Toe amputation (Surgical and medical procedures) | 1 | 1
Transurethral bladder resection (Surgical and medical procedures) | 1 | 0
Urethral repair (Surgical and medical procedures) | 1 | 0
Vertebra dislocation reduction (Surgical and medical procedures) | 1 | 0
Vertebroplasty (Surgical and medical procedures) | 1 | 0
(General disorders) | 4 | 2 — Details not available.
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0
Artery dissection (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 1
Hypovolaemic shock (Vascular disorders) | 2 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0
Leriche syndrome (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 10 | 2
Peripheral ischaemia (Vascular disorders) | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 2 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigation Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication. PIs may not publish single-site data until the main multi-site publication has occurred.